CLINICAL TRIAL: NCT06167785
Title: A Prospective, Multicenter, Phase II Trial to Evaluate the Efficacy of Zanubrutinib and Tislelizumab as Well as Standard of Care for the Treatment of Patients With Progressive Lymphoma Post Anti-CD19 CAR-T Cell Therapy
Brief Title: A Study to Evaluate Zanubrutinib and Tislelizumab in Progressive Lymphoma Post CAR-T
Acronym: ZeTA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OZUHN-024; NCT06919705 (obsolete NCT alias)
Record Dates: First submitted 2023-08-24; First posted 2023-12-13 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Large B-cell Lymphoma
MeSH Terms: interventions — tislelizumab; zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tislelizumab (Experimental): Tislelizumab 200mg intravenously every 3 weeks - initial safety run-in period
  Interventions: Drug: Tislelizumab
- Zanubrutinib (Experimental): Zanubrutinib 160 mg oral twice daily - initial safety run-in period
  Interventions: Drug: Zanubrutinib
- Tislelizumab + Zanubrutinib (Experimental): Tislelizumab 200mg intravenously day 1 of each cycle every 3 weeks
  * Zanubrutinib 160 mg oral twice daily starts day 1 of each cycle - expanded cohort
  Interventions: Drug: Tislelizumab + Zanubrutinib
- Standard of Care (No Intervention): Patients will receive standard of care, which is up to the investigator's discretion. This may include, but not limited to, palliative chemotherapy, steroids and/or radiation as deemed appropriate.

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg intravenously every 3 weeks
  Arms: Tislelizumab
Drug: Zanubrutinib — Zanubrutinib 160 mg oral twice daily
  Arms: Zanubrutinib
Drug: Tislelizumab + Zanubrutinib — Tislelizumab 200mg intravenously day 1 of each cycle every 3 weeks + Zanubrutinib 160 mg oral twice daily starts day 1 of each cycle
  Arms: Tislelizumab + Zanubrutinib

SUMMARY:
This is a phase ll study of participants with large B Cell lymphoma previously treated with anti-CD19 Chimeric antigen receptor (CAR-T) therapy. The purpose of the study is to to evaluate the efficacy of zanubrutinib and tislelizumab in patients with progressive lymphoma post anti-CD 19 CAR-T failure.

DETAILED DESCRIPTION:
Given that this group of patients is a heavily pre-treated group of individuals, the study will be broken into 2 distinct parts; an initial safety run-in period and an expanded cohort.

During both distinct parts of the study, patients meeting all the eligibility criteria except for the criteria specific to enrollment in the intervention arm, can be enrolled into the standard of care (SOC) arm.

Initial safety run-in period: intervention arm:

The initial safety run-in period will evaluate the tolerability and safety of tislelizumab or zanubrutinib monotherapy. In this initial phase, a total of 10 patients (5/ arm) will receive either zanubrutinib or tislelizumab monotherapy). Once the 10th patient has received 2 cycles of monotherapy, an early safety interim analysis will be complete to ensure the safety and tolerability of individual agents. These patients can continue to receive monotherapy until the results of the early safety interim analysis are known, at which point, if the study will move into the expanded cohort phase, these patients are eligible to receive the combination therapy.

Enrollment into the intervention arm will be paused after the enrollment of the 10th patient in the initial safety run-in period intervention arm, until it is determined the study will move into the expanded cohort phase. Enrollment of patients into the SOC arm can continue during this time.

Expanded cohort: intervention arm:

If monotherapy with tislelizumab and zanubrutinib are determined to be safe following the early safety interim analysis, then combination therapy will be explored in the expanded cohort. Patients will receive tislelizumab in combination with oral zanubrutinib. Patients that initially received monotherapy with tislelizumab or zanubrutinib, as part of the safety run in, will have the other drug added in for the remaining cycles. Patients will be allowed to continue in the study as long as they have acceptable toxicity profile and do not show disease progression, for up to a total of 34 cycles (~ 2 years) of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Able and willing to provide written informed consent and to comply with the study protocol
3. Radiologically measurable disease (≥ 1 nodal lesion > 2.0 cm in the longest diameter, and/or extranodal lesion > 1.0cm in the longest diameter)
4. Intervention arm: Radiological measureable disease per inclusion criterion #3 with more than one site of disease.
5. Relapse or refractory Large B cell Lymphoma post-CD19 directed CAR-T cell therapy within 6 weeks prior to enrollment (histological confirmation highly recommended although not mandatory)
6. Intervention arm: Hemoglobin ≥ 80 g/L at screening*
7. Intervention arm: Platelet count ≥ 50 x 109/L at screening*
8. Intervention arm: Neutrophil count ≥ 1.0 x 109/L at screening*
9. Intervention arm: performance status ≤ 2 at screening
10. AST and ALT < 2.5 x upper limit of normal (ULN) at screening
11. Serum total bilirubin < 1.5 x ULN, or < 3 x ULN in patients with documented Gilberts syndrome at screening
12. Creatinine clearance ≥ 30 mL/min as estimated by Cockcroft-gault equation at screening * Counts can be supported with growth factors or transfusions as per standard transfusion protocols

Exclusion Criteria:

1. Life expectancy < 30 days at the time of enrollment
2. Prior exposure to bruton tyrosine kinase (BTK) or Programmed cell death (PD)-1 inhibitor at any time prior to enrollment
3. Prior anaphylactic reaction to monoclonal antibody therapy at any time prior to enrollment
4. On higher than physiologic doses (10mg daily) of prednisone daily at least 7 days prior to initiation of trial treatment
5. Uncontrolled autoimmune disease
6. Known active central nervous system (CNS) involvement disease
7. History of prior allogeneic transplant or organ transplant
8. Active bleeding or history of bleeding diathesis including, but not limited to,

   * History of severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention
   * History of stroke or intracranial hemorrhage within 180 days before first dose of study drug
9. Difficulty with or unable to swallow oral medication, or known conditions that would significantly affect gastrointestinal function that would limit absorption of oral medication
10. History of chronic or active, uncontrolled bacterial, viral or fungal infection; human T- cell lymphotropic virus type 1 seropositive status.
11. Serologic status reflecting active viral hepatitis B or C infection as follows: (a) presence of hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Patients with presence of HBcAb, but absence of HBsAg, are eligible if hepatitis B virus (HBV) deoxyribonucleic acid (DNA) is undetectable (< 20IU), and if they are willing to be on appropriate prophylaxis and undergo monitoring for HBV reactivation if clinically indicated.

    (b) Presence of hepatitis C virus (HCV) antibody. Patients with presence of HCV antibody are eligible if HCV ribonucleaic acid (RNA) is undetectable.
12. Individuals with known active human immunodeficiency (HIV) infection are eligible if CD4 and viral titres are controlled
13. Any serious intercurrent illness, life threatening condition, organ system dysfunction including:

    * (1) Clinically significant cardiovascular including:

      1. prolonged QTc > 480ms,
      2. history of Mobitz II second degree or third degree heart block without a permanent pacemaker in situ,
      3. uncontrolled hypertension as indicated by a minimum of 2 consecutive blood pressure reading on 2 separate occasions showing systolic blood pressure (BP) > 170 mmHg and/or diastolic BP > 105mmHg at screening,
      4. uncontrolled or history of symptomatic arrhythmias (ie. sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes),
      5. congestive heart failure or NYHA class ≥ 3,
      6. myocardial infarction within 6 months prior to enrollment;
    * (2) History of significant cerebrovascular events including stroke or intracranial hemorrhage within 6 months prior to enrollment
    * (3) History of interstitial lung disease or non-infectious pneumonitis (excluding radiation induced), or severe/ debilitating pulmonary disease prior to enrollment
14. History of other active malignancies within 2 years prior to enrollment, with the exception of adequately treated in-situ carcinoma of cervix; localized basal cell or squamous cell carcinoma of skin; or previous malignancy confined and treated locally (surgery or other modality) with curative intent.
15. Female patients of childbearing potential must practice highly effective methods (Section 6.7.1.1) of contraception initiated prior to first dose of study drug, for the duration of the study, and for ≥ 90 days after the last dose of zanubrutinib or tislelizumab
16. Male patients are eligible if vasectomized or if they agree to the use of barrier contraception with highly effective methods during the study treatment period and for ≥ 90 days after the last dose of zanubrutinib or tislelizumab.
17. Major surgery within 4 weeks of the first dose of study drug
18. Vaccination with a live vaccine within 28 days prior to the first dose of study drug
19. Patient requires treatment with warfarin or other vitamin K antagonists
20. Severe or debilitating pulmonary disease (dyspnea at rest, significant shortness of breath, congestive obstructive pulmonary disease).
21. History of interstitial lung disease or noninfectious pneumonitis, except for those induced by radiation therapy.
22. Active and symptomatic fungal, bacterial, and/or viral infection; human T-cell lymphotropic virus type 1 seropositive status.
23. Any illness or condition that in the opinion of the investigator may affect safety of treatment or evaluation of any study endpoint.
24. Active autoimmune diseases or history of severe autoimmune diseases; these include but are not limited to a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis, systemic lupus erythematosus, rheumatoid arthritis, connective tissue diseases, scleroderma, inflammatory bowel disease, Crohn's disease, ulcerative colitis, autoimmune hepatitis, toxic epidermal necrolysis, Stevens-Johnson syndrome, or clinically manifest antiphospholipid syndrome. Note: Subjects are permitted to enroll if they have vitiligo, eczema, type I diabetes mellitus, or endocrine deficiencies, including thyroiditis managed with replacement hormones including physiologic doses of corticosteroids. Subjects with Sjögren's syndrome and psoriasis controlled with topical medication and subjects with positive serology, such as antinuclear antibodies or antithyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
25. A condition requiring systemic treatment with either corticosteroids (> 20 mg daily prednisone or equivalent) or other immunosuppressive medications within 14 days of study drug administration, except for primary central nervous system lymphoma (PCNSL) and secondary central nervous system lymphoma (SCNSL). Note: adrenal replacement doses ≤ 20 mg daily prednisone or equivalents are permitted in the absence of active autoimmune disease; subjects are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).
26. Major surgery in the past 4 weeks prior to the first day of screening.
27. Intervention arm: Live vaccines within 28 days of screening
28. Patients with contraindications for zanubrutinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
determine the best overall response rate (ORR) | 2 years
  To determine the best overall response rate (ORR) of the combination of zanubrutinib and tislelizumab as well as standard of care in patients previously treated with anti-CD19 CAR-T cell therapy. The best ORR is defined as the proportion of patients with a complete response (CR) or a partial response (PR) during the study, as determined by the investigator using Lugano 2014 criteria.

SECONDARY OUTCOMES:
Duration of response (DOR) | 2 years
  DOR is defined as the time from the first occurrence of a documented objective response (CR or PR) to disease progression or relapse, as determined by the investigator using Lugano 2014 criteria, or death from any cause, whichever occurs first
Progression free survival (PFS) | 2 years
  PFS is defined as the date of enrollment until disease progression, relapse or death from any cause
Event free survival (EFS) | 2 years
  EFS is defined as the date of enrollment until disease progression, relapse, death, or discontinuation of treatment for one of three reasons: toxicity, patient preference, initiation of new treatment without documented progression
Overall survival (OS) | 2 years
  OS is define as the date of enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: John Kuruvilla, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network (UHN), Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No